CLINICAL TRIAL: NCT05645263
Title: The Randomized Controlled Trial of Coca-cola's Clinical Effects on Gastric Phytobezoars
Brief Title: Coca-cola's Clinical Effects on Gastric Phytobezoars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhanglingyun，MD, Principal Investigator, The Affiliated Hospital of Qingdao University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: zhanglingyunzhanglingyun
Record Dates: First submitted 2022-11-22; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Bezoars
Keywords: RCT; Bezoars; Cola; lithotripsy; Gastroscopy
MeSH Terms: conditions — Bezoars

STUDY DESIGN:
Intervention Model Description: All patients were divided into 3 groups according to bezoar formation time combined with the willing of the patients. Patients whose phytobezoar formation time was less than a week in Group 1 , phytobezoar formation time between 1week and 2 weeks in Group2 , phytobezoar formation time longer than 2 weeks in Group 3. Every group was subdivided into intervention and control group according to whether Coco-cola was dieted.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor don't know which group the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cola 1（3d） (Experimental): The patients in intervention group 1 dieted Coca-cola to treat gastric phytobezoars, 250ml-500ml/2 h till to sleeping time according to the health conditions and life habits. Pay more attention to the stools and assess if the bezoars had excreted. The dieting Coca-cola period is 3 days.The patients will go through an endoscopy once the Coca-cola dieting therapy is over.
  Interventions: Other: dieting Coca-cola
- Cola 2（5d） (Experimental): The patients in intervention group 2 dieted Coca-cola to treat gastric phytobezoars, 250ml-500ml/2 h till to sleeping time according to the health conditions and life habits. Pay more attention to the stools and assess if the bezoars had excreted. The dieting Coca-cola period is 5 days. The patients will go through an endoscopy once the Coca-cola dieting therapy is over.
  Interventions: Other: dieting Coca-cola
- Cola 3（7d） (Experimental): The patients in intervention group 3 dieted Coca-cola to treat gastric phytobezoars, 250ml-500ml/2 h till to sleeping time according to the health conditions and life habits. Pay more attention to the stools and assess if the bezoars had excreted. The dieting Coca-cola period is 7 days. The patients will go through an endoscopy once the Coco-cola dieting therapy is over.
  Interventions: Other: dieting Coca-cola
- Fragmentation 1 (No Intervention): The patients who chose emergently endoscopic fragmentation was enrolled in control group 1. All patients endorsed the informed consent paper, no diet for at least 4 hours, no drink for 2 hours and bring the medical records before endoscopy and go on a mechanical fragmentation through gastroendoscopy
- Fragmentation 2 (No Intervention): The patients who chose emergently endoscopic fragmentation was enrolled in control group 2. All patients endorsed the informed consent paper, no diet for at least 4 hours, no drink for 2 hours and bring the medical records before endoscopy and go on a mechanical fragmentation through gastroendoscopy
- Fragmentation 3 (No Intervention): The patients who chose emergently endoscopic fragmentation was enrolled in controlled Group 3. All patients endorsed the informed consent paper, no diet for at least 4 hours, no drink for 2 hours and bring the medical records before endoscopy and go on a mechanical fragmentation through gastroendoscopy

INTERVENTIONS:
Other: dieting Coca-cola — The patients all dieted Coco-cola to treat gastric phytobezoars, 250ml-500ml/2 h till to sleeping time according to the health conditions and life habits. Pay more attention to the stools and assess if the bezoars had excreted. The dieting Coco-cola period of group A is 3 days, group B is 5 days and group C is 7 days.
  Arms: Cola 1（3d）; Cola 2（5d）; Cola 3（7d）

SUMMARY:
Consecutive patients suffering from gastric phytobezoars were divided into 3 groups (Group 1, Group 2 and Group 3) according to the phytobezoars' formation time and each group was further subdivided into control and intervention group according to whether Coca-Cola was admitted. All patients in intervention group dieted Coca-Cola whereas patients in control group refused to drink Coca-Cola and had willing to receive the emergently gastric fragmentation.

DETAILED DESCRIPTION:
Consecutive patients were enrolled and were divided into Group 1(the formation time of phytobezoars was less than 7 days), Group 2(the formation time of phytobezoars was from 7 days to 14 days) and Group 3 (the formation time of phytobezoars was more than 14 days) according to the formation time of phytobezoars and each group was subdivided into control group (who refused to diet Coca-Cola and chose emergent fragmentation with gastroscopy) and intervention Group (who had a willing to diet Coca-Cola) from 1st Jan, 2017 to 1st Dec 2021. The current protocol was approved by the Medical Ethics Committee of the Affiliated Hospital of Qingdao University (QYFYWZLL 26293). The patients in intervention group all dieted Coca-Cola to treat gastric phytobezoars, 250ml-500ml/2 h till to sleeping time according to personal health conditions and life habits. Pay more attention to the stools and assess if the bezoars had excreted. The Coca-Cola dieting period of intervention group 1 was 3 days, intervention group 2 was 5 days and intervention group 3 was 7 days. The patients would go through an endoscopy once the Coca-Cola dieting therapy was over. The patients who chose emergently endoscopic fragmentation was enrolled in control Group. All patients endorsed the digital informed consent and bring the medical records before endoscopy. Statistical analysis was performed with SPSS version 22(IBM, Inc. Armonk, NY, USA). ANOVA or independent samples t-test was used for analysis of continuous variables. P < 0.05 was taken as statistical meaning.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by abdominal CT or gastroscope;
* years older than 12;
* no contraindications;
* have willingness to diet Caco-cola to treat gastric bezoars;
* choose the emergent endoscopy whose bezoar formation time are more than 2 weeks;

Exclusion Criteria:

* Gastroscopy contraindications;
* choose the emergent endoscopy whose bezoar formation time are shorter than 2 weeks;
* years younger than 12 years;

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Dissolution rate | up to 48 months
  All the patients will go through a repeated endoscopy to ascertain if the phytobezoars has disappeared or shrinked and record the findings
Medical expense | up to 48 months
  The medical expense of each patient was added together and compared among the groups
Operation time | up to 48 months
  The operation time of each patient was recorded and compared among the groups
Gastric ulcer rate | up to 48 months
  All the patients will go through a repeated endoscopy to ascertain if there was ulcers located in the stomach and record the findings

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, PHD, Study Chair — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
There isn't a plan to make individual participant data available to other researchers